CLINICAL TRIAL: NCT01119040
Title: Prospective Evaluation of NOTES PEG "Rescue"
Brief Title: Prospective Evaluation of NOTES (Natural Orifice Translumenal Endoscopic Surgery) PEG "Rescue"
Acronym: PEGRescue
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Jeffrey Marks, MD, Principal Investigator, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-07-23
Record Dates: First submitted 2010-05-06; First posted 2010-05-07 (Estimated); Results first posted 2012-12-03 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2014-12

CONDITIONS: Malnutrition
Keywords: Dislodged PEG tube; NOTES
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NOTES PEG Rescue (Experimental): A new way of performing surgery is called Natural Orifice Translumenal Endoscopic Surgery, or NOTES, for short. NOTES may allow surgeons to perform abdominal surgery without any skin incisions. By using natural openings in the body, like the mouth, surgeons can enter the stomach with a tube instead of the traditional method of making an incision in the skin of the abdomen.
  Interventions: Procedure: Natural Orifice Translumenal Endoscopic Surgery

INTERVENTIONS:
Procedure: Natural Orifice Translumenal Endoscopic Surgery — Natural Orifice Translumenal Endoscopic Surgery (NOTES) procedures involve transmural passage of flexible endoscopes introduced via a natural orifice whereby permitting access to the peritoneal cavity while avoiding skin incisions. No clear indication due to a number of physiologic, microbiologic, immunologic, and technical limitations. The concept of NOTES PEG "Rescue" in the setting of a dislodged naïve PEG tube may spare individual patients the physiologic stress of traditional surgery while concomitantly providing a natural segue to further study the NOTES platform in the human setting. PEG "Rescue" may represent a unique, practical, and empowering application of the burgeoning experience of natural orifice translumenal endoscopic surgery.
  Other Names: NOTES

SUMMARY:
The purpose of this study is to determine:

1. Utility of urgent upper endoscopy in setting of dislodges (percutaneous endoscopic gastrostomy) PEG tube.
2. Feasibility of replacing naive PEG tubes with Natural Orifice Translumenal Endoscopic Surgery (NOTES) in lieu of traditional surgical methods.
3. Efficacy of replacing naive PEG tubes with NOTES in lieu of traditional surgical methods.

DETAILED DESCRIPTION:
1. Utility of Urgent Upper Endoscopy in Setting of Naïve Dislodged PEG Tubes as defined by:

   * Percentage of Open vs. Closed Gastrotomy upon urgent endoscopy
   * Presence of Incidental Pathology noted on Endoscopy
   * Complications of Urgent Endoscopy
   * Time of Procedure
2. Technical Feasibility of the NOTES procedure determined by:

   * Number of Successful/Failed PEG Placements
   * Number of Patients Requiring intra-operative conversion to laparotomy or laparoscopic procedure
   * Time to Complete Procedure
   * Presence or absence of post-procedural contrast extravasation on completion contrast radiographic study
3. Efficacy of NOTES PEG Rescue compared to historical controls as characterized by the following post-operative criteria:

   * Number of Patients Requiring Subsequent Medical or Surgical Treatment for Intra-Abdominal Abscess
   * Number of Patients Requiring Subsequent Medical or Surgical Wound Infection within 30 post-op days
   * Post-Operative CT or Operative Findings consistent with abscess confirmed by culture positive drainage, aspiration
   * Intra-Operative or Post-Operative Red Blood Cell Transfusion
   * Length of Stay
   * Antibiotics > 24h Post-Op
   * 30 day Re-Admission
   * Mortality

ELIGIBILITY:
Inclusion Criteria: Patients must meet ALL of the following criteria

* For prospective candidates, an initial attempt to pass a balloon tipped foley catheter through the external cutaneous tract into the stomach will be performed. It will then be followed by radiographic contrast study to evaluate for extravasation of contrast into the peritoneal cavity. If contrast is extravasated, this will be potential candidate for inclusion. If the foley catheter is unable to be passed through the cutaneous tract, that will also be considered someone for inclusion as this patient will still require an operative confirmation of the patency of the gastrotomy.
* For retrospective candidates, intra-operative confirmation of dislodged tube as reported in the medical record.
* The patient must demonstrate pre-operative hemodynamic and respiratory stability
* No overwhelming medical co-morbidities prohibitive of surgery
* Subject is 18 years of age or older
* Subject or subject's legal decision-making proxy agrees to participate, fully understands and signs the informed consent form

Exclusion Criteria: Patients must not meet ANY of the following criteria:

* Esophageal stricture prohibiting passage of an endoscope
* Any contraindication to surgery
* Pregnancy or actively breastfeeding women
* Evidence of active bowel obstruction
* Synchronous acute abdominal pathology warranting incision-based surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-11; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Marks, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Result] Marks JM, Ponsky JL, Pearl JP, McGee MF. PEG "Rescue": a practical NOTES technique. Surg Endosc. 2007 May;21(5):816-9. doi: 10.1007/s00464-007-9361-2. Epub 2007 Apr 3. PMID 17404790

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at University Hospitals Case medical Center between November 2007 and July 2010.
Groups:
- NOTES "PEG Rescue": Natural Orifice Translumenal Endoscopic Surgery (NOTES) procedures involve transmural passage of flexible endoscopes introduced via a natural orifice whereby permitting access to the peritoneal cavity while avoiding skin incisions.
Period: Overall Study
Arm/Group | NOTES "PEG Rescue"
Started | 1
Completed | 0
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Peg Rescue: Peg Rescue with NOTES in lieu of traditional surgical methods for dislodged PEG tubes.
Arm/Group | Peg Rescue
Number analyzed (Participants) | 1
Age, Customized [Number; unit: Participants]
  Over the age of 18 yrs | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1
number of days to assure leak-proof gastrocutaneous tract [Number; unit: Days] — Following initial placement of a PEG tube, a variable number of days is required to assure a leak-proof gastrocutaneous tract formed between the adherent stomach serosa and the parietal peritoneum of the anterior wall. In well-nourished, healthy individuals free of wound-healing impairment, a robust gastrotomy track is typically formed within 2 to 4 weeks. For PEG tubes dislodged in the first two weeks post-operatively, the risk of an incompletely formed gastrocutaneous fistula track prompts concern for intra-abdominal leakage from gastrotomy.
  Days | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Replacements of Dislodged PEG Tubes With NOTES Procedures in Lieu of Traditional Surgical Methods.
Description: Successful replacement will be determined via the number of patients requiring conversion from NOTES PEG rescue to conventional incision-based surgery.
Time Frame: 30 day follow-up
Population: Only 1 subject due to low accrual
Measure: Number; unit: participants
Groups:
- NOTES PEG Rescue: Natural Orifice Translumenal Endoscopic Surgery (NOTES) procedures involve transmural passage of flexible endoscopes introduced via a natural orifice whereby permitting access to the peritoneal cavity while avoiding skin incisions.
Arm/Group | NOTES PEG Rescue
Number analyzed (Participants) | 1
participants | 1

ADVERSE EVENTS:
Groups:
- NOTES PEG Rescue: Peg Rescue with NOTES in lieu of traditional surgical methods for dislodged PEG tubes.
Arm/Group | NOTES PEG Rescue
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Study terminated early due to difficulty with patient accrual due to lack of patient population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No